CLINICAL TRIAL: NCT02592135
Title: High Sensitivity cTnT Rules Out Cardiac Insufficiency Trial (TACIT)
Acronym: TACIT
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Vanderbilt University (Other); Wayne State University (Other); University of Cincinnati (Other)
Responsible Party: Principal Investigator, PETER S PANG, Associate Professor, Indiana University
Other Study IDs: INEMER-0001
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Heart Failure
Keywords: Acute Cardiac Insufficiency; Acute Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum specimens for bio marker analysis
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: hsTnT level — hsTnT and NTproBNP levels at baseline and baseline plus 3 hours.

SUMMARY:
The purpose of this study is to better understand myocardial injury in AHF. Secondary analyses demonstrate the prognostic significance of troponin release. The absence of such release has been associated with less risk. Whether measurement of high sensitivity TnT may enable emergency physicians to better risk stratify acute heart failure patients remains to be determined. This study will help us to better understand the prognostic value of absent or low hsTnT values in the emergency department setting. In addition, we will also test the STRATIFY decision rule; a risk score.

DETAILED DESCRIPTION:
Hospitalization for acute heart failure (AHF) results in a high rate of post-discharge mortality and re-admissions, as well as high financial costs. Reducing 30-day re-admissions after AHF hospitalization is a major national quality goal intended to both improve patient outcomes and reduce costs.

Approximately 85% of emergency department (ED) patients with AHF are hospitalized, and 800,000 of the 1,000,000 hospitalizations for HF originate from the ED, highlighting the critical role of the ED. Even a single digit percentage (i.e. 5%) decrease in the number of AHF admissions would equate to an estimated 40,000 fewer hospitalizations.

Why are so many AHF patients hospitalized? AHF patients have a high post-discharge event rate. Emergency physicians have a low risk tolerance. When both are combined, most patients are admitted. The absence of risk scores for the ED setting compounds the problem. Most risk scores were developed in the hospital. As hospitalization may affect the outcomes of patients, whether these risk scores apply to the ED setting is unknown. As a result, which patients are at lower risk in the ED has not been well-studied. Further, absence of high-risk features does not necessarily equal absolute low morbidity or mortality, though such patients are likely at lower risk. In the absence of a risk score, clinical judgment is a poor substitute and often fails to identify patients at high risk, such that those discharged from the ED may be at equal or greater risk for death than hospitalized patients. Thus, the difficulty of identifying low risk, combined with the inherent high morbidity and mortality of AHF, leads to a disproportionate number of hospitalizations.

Over a decade ago, the Agency for Healthcare Research and Policy Guidelines suggested that up to 50% of AHF patients were potential candidates for ED discharge or observation unit management. Furthermore, nearly half of all patients hospitalized for AHF present with lower-risk features such as high blood pressure (> 140mmHg) and a BNP < 1000 pg/mL. If low or lower risk ED patients with HF could be accurately identified, perhaps a greater proportion of patients with AHF could be safely discharged or observed briefly prior to discharge.

Study Rationale: With this pilot study, we will generate the necessary and sufficient pilot data to inform the design of a definitive trial to test whether identification of low risk acute heart failure (AHF) patients with negative serial high-sensitivity troponin T (hsTnT) in the ED may be safely discharged home or observed briefly in observation status.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥21 years old
2. Patient diagnosed with acute heart failure (AHF) by the treating physician.
3. Patient has received IV loop diuretic or vasodilator therapy (by any route) for AHF
4. Provide informed written consent
5. SBP > 100mmHg

Exclusion Criteria:

1. Life expectancy ≤6 months
2. Shock of any kind or use or planned use of inotropes (dobutamine, dopamine, milrinone) or vasopressors. Any form of vasodilator is allowed.
3. Fever > 101.5
4. Presumed ACS as primary reason for presentation or ACS within 30 days. Patients with troponin release outside of ACS (Type 2 MI) may be included
5. AF with RVR > 130bpm at any time requiring medical intervention
6. History of transplant of any kind or VAD patient
7. ESRD requiring dialysis
8. Involved in any investigational trial (observational study where there is no intervention is allowed)
9. Currently under treatment for cancer of any kind
10. Alcohol or other substance abuse
11. Any patient whom the investigator deems would be difficult to obtain follow-up

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the Emergency Department (ED) with signs and symptoms of AHF
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-12-21 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
A composite of all cause mortality and re-hospitalization, including ED re-visits | 90 days
  Have increased the follow up from 30 to 90 days. Will also analyze for 30 days

SECONDARY OUTCOMES:
Days alive and out of hospital | 90 days
  Will also analyze for 30 days
Cardiovascular specific re-hospitalization and ED revisits | 90 days
  Will also analyze for 30 days
Hierarchial Adverse Events Model (STRATIFY Risk Score) | 90 days
  Will also analyze for 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Pang, MD, Principal Investigator — Indiana University
Locations (5):
- United States (5):
  - Eskenazi Health, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Detroit Receiving Hospital, Detroit, Michigan
  - University of Cincinnati, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pang PS, Fermann GJ, Hunter BR, Levy PD, Lane KA, Li X, Cole M, Collins SP. TACIT (High Sensitivity Troponin T Rules Out Acute Cardiac Insufficiency Trial). Circ Heart Fail. 2019 Jul;12(7):e005931. doi: 10.1161/CIRCHEARTFAILURE.119.005931. Epub 2019 Jul 10. PMID 31288565